CLINICAL TRIAL: NCT02136589
Title: Effect of Non-steroid Anti-inflammatory Drug on Travoprost-induced Conjunctival Hyperemia and Intraocular Pressure Reduction in Normal Eyes
Brief Title: Effect of NSAID on Travoprost-induced Conjunctival Hyperemia and IOP Reduction in Normal Eyes
Acronym: ENTICHIR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tokyo University (Other)
Responsible Party: Principal Investigator, Makoto Aihara, Associate Professor, Tokyo University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CS-097
Record Dates: First submitted 2011-07-20; First posted 2014-05-13 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Hyperemia; Intraocular Pressure
MeSH Terms: conditions — Hyperemia | interventions — Diclofenac; Travoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dicrofenac (Experimental)
  Interventions: Drug: dicrofenac and travoprost

INTERVENTIONS:
Drug: dicrofenac and travoprost — dicrofenac drop 3 times a day travoprost 0.005% once daily

SUMMARY:
PG-analogues induce hyperemia as one of side effects in addition to IOP reduction.

IOP reduction is caused by direct FP receptor stimulation, but the cause of hyperemia is not clarified.

Because FP receptor stimulation induce intrinsic production of PGs, hyperemia or IOP reduction may be due to secondary induced PGs.

Thus, pretreatment with NSAID may affect the PG-analogue induced hyperemia or IOP reduction.

ELIGIBILITY:
Inclusion Criteria:

1. normal healthy eye
2. not applicable for IOP level
3. not wearing contact lenses
4. not applicable for the presence of the ocular surface diseases in case the treatment was not needed

Exclusion Criteria:

1. the eyes with chronic or recurrent uveitis, scleritis, corneal herpes infection
2. the eyes with the history of trauma, intraocular surgery, or Laser surgery within 6 months
3. the eyes with difficulty for the measurement of IOP with the applanation tonometer
4. the subjects with the allergy for PG-analogues or benzalkonium chloride
5. the subjects using the eyedrops excluding those in this study
6. the subjects treated with oral carbonic anhydrase inhibitor
7. the subject with Sjogren syndrome
8. the subjects who can not drop periodically
9. the subjects with the advanced glaucoma or the terminal stage of glaucoma
10. the subjects with the severe ocular complications

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
IOP reduction | 1 day
  effect of NSAID on IOP reduction by travoprost